CLINICAL TRIAL: NCT06757270
Title: Efficacy of Aleo Vera Use in Prevention and Treatment of Chemotherapy-Induced Oral Mucositis in a Group of Egyptian Children with Acute Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FDASU-EecIM 022203
Record Dates: First submitted 2024-12-17; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-03

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alovera experminted arm (Experimental)
  Interventions: Other: Second arm: Using aleovera for Prevention and Treatment of Chemotherapy-Induced Oral Mucositis
- second group (No Intervention)

INTERVENTIONS:
Other: Second arm: Using aleovera for Prevention and Treatment of Chemotherapy-Induced Oral Mucositis — Second arm : aleovera 3 times daily after brushing teeth
  Arms: Alovera experminted arm

SUMMARY:
evaluatation the efficacy of Aleovera in prevention and treatment of chemotherapy-induced oral mucositis in children suffering from acute leukemia in terms of appearance and severity

ELIGIBILITY:
Inclusion criteria

1. Patients suffering from Acute leukemia( Acute Lymphocytic Leukemia ).
2. Patients scheduled for chemotherapy treatment.
3. Patients who range from 3 to 13 years old.
4. Patients with no history of any chemotherapy or radiotherapy. 5 -Both sexes Exclusion Criteria

1-Patients scheduled for radiotherapy treatment . 2-Existence of any signs or symptoms of oral mucositis. 3-Unwilling to participation in the study 4- Patients with any other systemic diseases or other neoplasms.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Prevention of oral mucositis | 2 months
  Assessment the efficacy of aleo vera gel on prevention of chemotherapy-induced oral mucositis through application the gel 3 times daily then patients were assessed daily in terms of appearance and severity of oral mucositis according WHO grading system.
  The World Health Organization (WHO) mucositis scale is used to grade the severity of oral mucositis.
  Grade 0: No mucositis Grade 1: Soreness/erythema only. Grade 2: Erythema, and ulcers. Able to tolerate solids. Grade 3: Unable to tolerate solids but able to tolerate liquids. Grade 4: Unable to tolerate solids or liquids. Oral alimentation is not possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
after analysis of my results, if be with value i will share